CLINICAL TRIAL: NCT05424016
Title: Efficacy of Propranolol for the Treatment of Central Nervous System Hemangioblastomas in Von Hippel-Lindau Disease: a Randomized Controlled Clinical Trial
Brief Title: Propranolol and Von Hippel-Lindau Disease
Acronym: PRO-HEB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Générale des Equipements et Produits de Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210075; 2022-001174-54 (EudraCT Number)
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Hemangioblastoma of CNS; Von Hippel-Lindau Disease
Keywords: hemangioblastomas; Propranolol; Von Hippel-Lindau,; MRI
MeSH Terms: conditions — von Hippel-Lindau Disease; Hemangioblastoma | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: open-label, randomized, controlled trial with 2 parallel arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Patients with no contraindications will be included and randomized to receive propranolol orally for 24 months
  Interventions: Drug: Propranolol
- control arm (Other): Patient included with a routine follow-up
  Interventions: Other: follow-up

INTERVENTIONS:
Drug: Propranolol — 120 mg/d propranolol started in a progressive way (with control of Blood Pressure and heart rate during the consultations) neurosurgical consultation and an MRI every six months
  Arms: Experimental arm
Other: follow-up — routine follow-up (neurosurgical consultation and an MRI every six months)
  Arms: control arm

SUMMARY:
Propranolol (beta-blocker), is successfully used for the treatment of infantile hemangiomas, the most common vascular tumor of newborns. The mechanism is related to its anti-angiogenetic and pro-apoptotic effects. Recently, in vitro studies demonstrated that propranolol decreased the expression of target genes of the HIF (hypoxia-inducible factor, of which the VHL gene is the main regulator) pathway in hemangioblastoma cells and affected their viability. The efficacy of propranolol (stabilization of all HB and decrease in serum VEGF levels) was demonstrated in a phase III study, but only in retinal BHs . The only study that evaluated the effect of propranolol on CNS HB was retrospective and involved a limited number of patients. Nevertheless, it showed a decrease in the growth rate of HBs. The investigator therefore propose to carry out a randomized controlled trial to study the effect of propranolol on the growth of CNS HB in patients with VHL disease (von Hippel-Lindau).

The hypothesis of the present work is the following: the use of propranolol in VHL patients with CNS HB allows to decrease and/or slow down the tumor growth.

DETAILED DESCRIPTION:
'Von Hippel-Lindau disease (VHL) is a familial syndrome, autosomal dominant, of predisposition to cancer, associating malignant tumors (renal carcinomas, neuroendocrine tumors of the pancreas), or benign tumors (retinal hemangioblastomas (HB), cerebellar, spinal cord, endolymphatic sac tumors and pheochromocytomas, which is a consequence of a high-penetrance mutations in the VHL tumor-suppression gene. A patient with multiple HB may require multiple interventions, which may leave progressively severe neurological sequelae. Several drug treatments (interferon, tyrosine kinase inhibitors, anti-angiogenic agents) have been proposed and tested as alternatives to surgery or to delay it. None of these studies have demonstrated a favorable benefit-risk balance that would support the use of any of these treatments, which sometimes have major side effects, in routine practice. Propranolol (beta-blocker) is successfully used for the treatment of infantile hemangiomas, the most common vascular tumor of newborns. The mechanism is related to its anti-angiogenetic and pro-apoptotic effects. Recently, in vitro studies demonstrated that propranolol decreased the expression of target genes of the HIF (hypoxia-inducible factor, of which the VHL gene is the main regulator) pathway in hemangioblastoma cells and affected their viability. The efficacy of propranolol (stabilization of all HB and decrease in serum VEGF levels) was demonstrated in a phase III study, but only in retinal HB. The only study that evaluated the effect of propranolol on CNS HB was retrospective and involved a limited number of patients. Nevertheless, it showed a decrease in the growth rate of HB. The investigator therefore propose to perform a randomized controlled trial to study the effect of propranolol on CNS HB growth in patients with VHL disease. Patients will be introduced to the study during a routine follow-up visit or during a telephone call by their neurosurgeon. Eligible patients who have signed the consent form will have a cardiology consultation to rule out a contraindication to the use of propranolol, prior to inclusion/randomization. If a contraindication is detected by the cardiologist, the patient will not be included in the study.

Patients without contraindications will then be included and randomized (1:1) to receive either oral propranolol (120 mg/d, started gradually (with BP and heart rate monitoring at visits) for 24 months or usual follow-up. Randomization will be stratified on the number of initial CNS HB (<5 or ≥5).

Initial imaging (MRI) workup (brain and spinal cord) will be performed, with mapping and measurements of CNS HB, initially present.

Clinical (every three months) and radiological follow-up every 6 months (MRI) or when new neurological symptoms appear. Tolerance and secondary endpoints will also be assessed during these follow-up visits. Patients will be followed up to 26 months post-randomization.

The primary endpoint will be assessed centrally by two neuroradiologists, blinded to the patient's treatment arm. The other radiological endpoints (edema, growth velocity, de novo HB occurrence) will also be assessed centrally, by the same neuroradiologists, blinded to the treatment arm.

During follow-up, the use of surgery will not be modified by the protocol, and will be left to the discretion of the physician in charge of the patient, according to current recommendations. Statistical analysis:

Randomization will be performed in a 1:1 ratio between the two groups. It will be stratified on the initial number of CNS HB (<5 or ≥5). Efficacy endpoint analyses will be performed on the intention-to-treat (ITT, all randomized patients) population, in which all patients will be analyzed according to the allocated group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* VHL patient with one or more hemangioblastomas of the central nervous system, none of which require urgent surgery (within 3 months)
* Patient with written consent to participate in the study
* Enrolled in a social security plan or beneficiary

Exclusion Criteria:

* Contraindication to the use of propranolol:
* chronic obstructive pulmonary disease and asthma,
* uncontrolled heart failure,
* 2nd and 3rd degree atrioventricular blocks,
* bradycardia (<50 beats/minute after 3 minutes of rest),
* Raynaud's phenomenon and peripheral arterial disorders,
* arterial hypotension,
* hypersensitivity to propranolol
* cardiogenic shock,
* Prinzmetal's angina,
* sinus disease (including sino-auricular block)
* untreated pheochromocytoma,
* history of anaphylactic reaction,
* in the context of primary and secondary prevention of digestive bleeding in cirrhotics: advanced liver failure with hyperbilirubinemia, massive ascites, hepatic encephalopathy
* predisposition to hypoglycemia (as after fasting or in case of abnormal response to hypoglycemia)
* metabolic acidosis
* Contraindication to MRI:
* claustrophobia,
* presence of a pace maker and other stimulators/implants
* ocular metallic foreign bodies,
* heart valves or ferromagnetic metal vascular clips
* Patients already on Propranolol or other beta blockers
* Patients under guardianship or conservatorship
* Pregnant or breastfeeding women - Woman with a medium-term pregnancy project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
total and individual hemangioblastomas' volume measured by MRI | 24 months
  Response to treatment at 24 months will be a binary variable (responder/non responder) using initial imaging data and 24-month post-randomization, assessed by two neuroradiologists, independently.
  On baseline imaging two types of CNS BHs will be defined and measured:
  "measurable" BHs whose largest diameter is ≥ 5 mm "Non-measurable" BHs whose largest diameter is < 5 mm For each patient the sum of the volumes of all measurable BHs in mm3 will be calculated initially and compared to this same sum at 24 months post-randomization.
  A patient will be as "responder" :
  The sum at 24 months remains stable Or regresses No HB identified as "non-measurable" initially has reached the "measurable" criterion No de novo HBs have appeared
  A patient will be as "non-responder":
  The sum at 24 months increases At least one HB identified as "non-measurable" initially has reached the "measurable" criterion At least one de novo HB appears The patient has required surgery during follow-up

SECONDARY OUTCOMES:
To compare the safety (tolerance) between the two treatment arms at 24 months post-randomization | 24 months
  To study safety (tolerability) of propranolol in VHL patients: All adverse events related to the use of Propanolol that occurred during the study will be collected, analyzed and compared between the two treatment arms
To Compare the growth rate of HB between the two treatment arms at 24 months post-randomization | 24 months
  To compare HB growth rate between the two treatment arms at 24 months post-randomization: HB growth rate will be measured on each MRI by two neuroradiologists, blinded to the randomization arm. It will be calculated in mm3 /month using the function available on the ITK-SNAP imaging software ( www.itksnap.org.) which allows an accurate measurement of the tumor volume (In case of disagreement a conciliation session will be organized). The growth rate is therefore obtained by dividing the change in volume by the number of months between the two MRIs
Compare the extent of peritumoral edema between the two treatment arms | 24 months
  To compare the extent of peritumoral edema between the two treatment arms: The size of peritumoral edema will be measured on each MRI by two neuroradiologists, blinded to the randomization arm
Compare the development of de novo lesions between the two treatment arms every 6 months | 24 months
  To compare the occurrence of de novo lesions between the two treatment arms: the number of de novo HBs will be specified for each patient at each follow-up MRI by two neuroradiologists, blinded to the randomization arm. A de novo HB is defined as the appearance during follow-up of a HB that did not exist on the initial imaging (or the transition from a non-measurable HB to a measurable state
Compare the angiogenic profile of BHs between the two groups every 6 months | 24 months
  To compare the angiogenic profile of BHs between the two groups by perfusion sequence with r-CBV measurement for each measurable and perfusion-studyable lesion (> 1cm)
Study the evolution of serum VEGF level under treatment at 12 and 24 months | 24 months
  To study the evolution of serum VEGF level under treatment: Determination of serum VEGF level at the beginning of the treatment and then at 12 and 24 months by a simple peripheral venous blood sample. (pg/ml)
Compare the number of patients requiring surgery between the two treatment arms | 24 months
  To compare the number of patients requiring surgery between the two treatment arms: The use of surgery will be recorded during patient follow-up (use/non-use). The need for surgery will be left to the discretion of the physician responsible for the patient's follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France